CLINICAL TRIAL: NCT07221188
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, 3-Arm Study to Investigate the Safety and Tolerability of Efimosfermin Alfa in Participants With Known or Suspected F2- or F3-Stage Metabolic Dysfunction-Associated Steatohepatitis (MASH) (ZENITH-2)
Brief Title: A Clinical Study to Investigate the Safety and Tolerability of Efimosfermin Alfa Injection in Participants With Known or Suspected F2- or F3-stage MASH
Acronym: ZENITH-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 306246; 2025-523674-16 (Other: EU CT Number)
Record Dates: First submitted 2025-10-15; First posted 2025-10-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Metabolic Dysfunction-Associated Steatohepatitis; efimosfermin alfa; Safety; Tolerability; Phase 3; ZENITH-2
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Efimosfermin Alfa Dose Level 1 (Experimental): Participants randomized to this group will receive Efimosfermin Alfa at dose level 1
  Interventions: Drug: Efimosfermin Alfa
- Efimosfermin Alfa Dose Level 2 (Experimental): Participants randomized to this group will receive Efimosfermin Alfa at dose level 2
  Interventions: Drug: Efimosfermin Alfa
- Placebo (Placebo Comparator): Participants randomized to this group will receive Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Efimosfermin Alfa — Efimosfermin Alfa will be administered
  Arms: Efimosfermin Alfa Dose Level 1; Efimosfermin Alfa Dose Level 2
Drug: Placebo — Placebo will be administered
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and tolerability of Efimosfermin Alfa for participants with known or suspected MASH with fibrosis consistent with stage F2 or F3.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to understand and sign a written informed consent form (ICF) that must be obtained prior to the initiation of study procedures
* Age >=18 through <=75 years at enrolment
* History or presence of 2 or more of the 5 components of metabolic syndrome per American Heart Association definition
* History or presence of known or suspected MASH

Exclusion Criteria:

* ALT or AST >=5 × upper limit of normal (ULN)
* Total bilirubin (BILI) >=1.3 milligram per deciliter (mg/dL). Individuals with documented Gilbert's syndrome may be enrolled if they experienced an isolated increase in total BILI of >=1.3 mg/dL and direct BILI is <=20% of total BILI; otherwise, the individual will be excluded.
* Serum albumin <=3.5 grams per deciliter (g/dL)
* International normalized ratio (INR) >=1.3 not due to therapeutic anticoagulation. Individuals receiving chronic anticoagulant treatment with higher INR values may be enrolled at the discretion of the Investigator and Study Medical Monitor.
* Alkaline phosphatase (ALP) >=2 × ULN
* Platelet (PLT) count <140 000 per (/) cubic millimeter (mm^3); individuals with a PLT count between 110,000/mm^3 and 140,000/mm^3 may be enrolled after discussion with the Study Medical Monitor
* Serum creatinine >=1.5 mg/dL or creatinine clearance <=60 milliliter (mL)/minute (min)/1.73 square meter by Chronic Kidney Disease Epidemiology Collaboration equation.
* HbA1c >=9.0%
* Model for End-Stage Liver Disease (MELD) 3.0 score >=12 unless the score is elevated in the absence of liver dysfunction (eg, Gilbert's syndrome)
* Phosphatidylethanol (PEth) >=80 nanogram per milliliter (ng/mL) at Screening
* Known co-infection with any of the following: a. Human immunodeficiency virus; b. Hepatitis B virus; c. Hepatitis C virus (HCV); d. Hepatitis D virus; or e. Hepatitis E virus.
* Chronic liver disease from any other cause including, but not limited to, alcoholic liver disease; evidence of portal hypertension; viral hepatitis, or any history or evidence of cirrhosis; or decompensated liver disease such as clinical ascites, bleeding gastroesophageal varices, hepatorenal syndrome, or hepatic encephalopathy prior to Screening or Day 1.
* Current or history of excessive alcohol intake for >=3 months within the 12-month period prior to Screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2028-03-24 (Estimated); Study Completion 2028-03-24 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) and TEAEs by severity | At Week 52
Number of participants with TEAEs leading to discontinuation and TEAEs leading to discontinuation by severity | At Week 52
Number of participants with Grade 3 and Grade 4 laboratory abnormalities | At Week 52

SECONDARY OUTCOMES:
Absolute Change from Baseline in enhanced liver fibrosis (ELF) score | Baseline (Day 1) and up to Week 52
  The ELF score will be calculated using a published algorithm combining the values of a set of extracellular matrix markers. The ELF score is used as a prognostic marker for disease progression: ELF score less than (<) 9.8: Low risk of progression, ELF score 9.8 to <11.3: Moderate risk of progression and ELF score greater than or equal to (>=) 11.3: High risk of progression.
Percent Change from Baseline in ELF score | Baseline (Day 1) and up to Week 52
  The ELF score will be calculated using a published algorithm combining the values of a set of extracellular matrix markers. The ELF score is used as a prognostic marker for disease progression: ELF score <9.8: Low risk of progression, ELF score 9.8 to <11.3: Moderate risk of progression and ELF score >=11.3: High risk of progression.
Number of participants achieving an improvement in ELF score greater than equal to 0.5 | At Week 52
  The ELF score will be calculated using a published algorithm combining the values of a set of extracellular matrix markers. The ELF score is used as a prognostic marker for disease progression: ELF score <9.8: Low risk of progression, ELF score 9.8 to <11.3: Moderate risk of progression and ELF score >=11.3: High risk of progression.
Absolute Change from Baseline in vibration-controlled transient elastography (VCTE)- liver stiffness measurement (LSM) scores | Baseline (Day 1) and up to Week 52
Percent Change from Baseline in VCTE- LSM scores | Baseline (Day 1) and up to Week 52
Number of participants achieving a change from Baseline in VCTE-LSM >=30 percentage (%) | Baseline (Day 1) and up to Week 52
Absolute Change from Baseline in magnetic resonance elastography (MRE) scores in the subset of participants | Baseline (Day 1) and up to Week 52
  MRE is a non-invasive imaging technique that combine magnetic resonance imaging (MRI) scanning with low-frequency mechanical vibrations to measure the stiffness of liver. MRE scores <2.5 is normal, 2.5 - 3.0 Normal or inflammation, 3.0 - 3.5 Stage 1-2 fibrosis, 3.5 - 4.0 Stage 2-3 fibrosis, 4.0 - 5.0 Stage 3-4 fibrosis and > 5.0 Stage 4 fibrosis.
Percent Change from Baseline in the subset of participants with magnetic resonance elastography (MRE) scores | Baseline (Day 1) and up to Week 52
  MRE is a non-invasive imaging technique that combine MRI scanning with low-frequency mechanical vibrations to measure the stiffness of liver. MRE scores <2.5 is normal, 2.5 - 3.0 Normal or inflammation, 3.0 - 3.5 Stage 1-2 fibrosis, 3.5 - 4.0 Stage 2-3 fibrosis, 4.0 - 5.0 Stage 3-4 fibrosis and > 5.0 Stage 4 fibrosis.
Absolute Change from Baseline in hepatic fat fraction (HFF) by magnetic resonance imaging (MRI)- derived proton density fat fraction (PDFF) | Baseline (Day 1) and up to Week 52
  HFF is the percentage of fat in the liver measured by MRI proton density fat fraction technique, which ranges from 0-75%. Greater than 5% is considered extra fat in the liver.
Percent Change from Baseline in HFF by MRI-PDFF | Baseline (Day 1) and up to Week 52
  HFF is the percentage of fat in the liver measured by MRI proton density fat fraction technique, which ranges from 0-75%. Greater than 5% is considered extra fat in the liver.
Absolute Change from Baseline in alanine aminotransferase (ALT) and aspartate aminotransferase (AST) (International units per liter) | Baseline (Day 1) and up to Week 52
Absolute Change from Baseline in ALT and AST ratio (ALT/AST) | Baseline (Day 1) and up to Week 52
Percent Change from Baseline in ALT and AST (International units per liter) | Baseline (Day 1) and up to Week 52
Percent Change from Baseline in ALT and AST ratio (ALT/AST) | Baseline (Day 1) and up to Week 52
Number of participants achieving ALT and HFF normalization | At Week 52
Number of participants achieving HFF less than equal to (<=) 5% | At Week 52
  HFF is the percentage of fat in the liver measured by MRI proton density fat fraction technique, which ranges from 0-75%. Less than or equal to 5% is considered normal (no significant fatty infiltration (steatosis) in the liver.
Change from Baseline in glycated hemoglobin (HbA1c) for participants with type 2 diabetes mellitus (T2DM) | Baseline (Day 1) and up to Week 52
Change from Baseline in body weight for all participants(kilograms) | Baseline (Day 1) and up to Week 52
Change from Baseline in fasting total cholesterol, low-density lipoprotein (LDL)-cholesterol, high-density lipoprotein (HDL)- cholesterol, and fasting triglycerides (Millimoles per liter) | Baseline (Day 1) and up to Week 52
Number of Participants with antidrug and anti-fibroblast growth factor 21 (FGF21) antibodies (ADA) at Week 52 | At Week 52
Maximum serum drug concentrations (Cmax) of efimosfermin alfa | Up to Week 52
Area under the serum concentration-time curve (AUC) of efimosfermin alfa | Up to Week 52
Average serum drug concentration (Cavg) of efimosfermin alfa | Up to Week 52
Serum concentration of study drug at the end of the dosing interval (Ctrough) of efimosfermin alfa | Up to Week 52
Exposure-response relationship for efimosfermin alfa | Baseline (Day 1) and up to Week 52
  To evaluate the correlation between pharmacokinetics (PK) derived from plasma concentrations, and biomarker responses, safety, and efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (5):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf